CLINICAL TRIAL: NCT01234740
Title: BAFETINIB-P1-GBM-01: A Pilot Study Using Intracerebral Microdialysis to Determine the Neuropharmacokinetics of Bafetinib in Patients With Recurrent Brain Tumors
Brief Title: Bafetinib in Treating Patients With Recurrent High-Grade Glioma or Brain Metastases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10134; NCI-2010-01963
Record Dates: First submitted 2010-09-28; First posted 2010-11-04 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Adult Anaplastic Astrocytoma; Adult Anaplastic Ependymoma; Adult Anaplastic Oligodendroglioma; Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Adult Mixed Glioma; Recurrent Adult Brain Tumor; Tumors Metastatic to Brain; Adult Anaplastic Oligoastrocytoma
Keywords: Los Angeles
MeSH Terms: conditions — Astrocytoma; Ependymoma; Oligodendroglioma; Glioblastoma; Gliosarcoma; Glioma; Brain Neoplasms | interventions — bafetinib; Microdialysis; Chromatography, Liquid; Mass Spectrometry; Blotting, Western; Immunohistochemistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients undergo intracerebral microdialysis during debulking craniotomy or stereotactic biopsy. Beginning 24 hours later, patients receive oral bafetinib twice daily for 1 day. Beginning at least 2 weeks after surgery, patients continue to receive oral bafetinib twice daily in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: bafetinib; Procedure: microdialysis; Other: pharmacological study; Other: liquid chromatography; Other: mass spectrometry; Other: laboratory biomarker analysis; Genetic: protein expression analysis; Genetic: western blotting; Other: immunohistochemistry staining method; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Drug: bafetinib — Given orally
  Other Names: dual Bcr-Abl/Lyn tyrosine kinase inhibitor INNO-406; INNO-406; NS-187
Procedure: microdialysis — Catheter placed intracerebrally during debulking craniotomy or stereotactic biopsy
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: liquid chromatography — Correlative studies
  Other Names: LC
Other: mass spectrometry — Correlative studies
Other: laboratory biomarker analysis — Correlative studies
Genetic: protein expression analysis — Correlative studies
Genetic: western blotting — Correlative studies
  Other Names: Blotting, Western; Western Blot
Other: immunohistochemistry staining method — Correlative studies
  Other Names: immunohistochemistry
Procedure: therapeutic conventional surgery — debulking craniotomy

SUMMARY:
RATIONALE: Bafetinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This clinical trial studies bafetinib in treating patients with recurrent high-grade glioma or brain metastases.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the neuropharmacokinetics (nPK) and systemic levels of bafetinib in patients with recurrent malignant brain tumors.

SECONDARY OBJECTIVES:

I. To investigate the intrapatient variability of nPK parameters as assessed by intracerebral microdialysis.

II. To document the toxicity of bafetinib in this cohort of patients. III. To describe the response rate, progression-free survival, and overall survival in patients with malignant brain tumors treated with bafetinib.

IV. To assess for the expression of Lyn and Fyn kinases and phosphorylation status in pre-treatment tumor samples.

OUTLINE:Patients undergo intracerebral microdialysis during debulking craniotomy or stereotactic biopsy. Beginning 24 hours later, patients receive oral bafetinib twice daily for 1 day. Beginning at least 2 weeks after craniotomy or 1 week after biopsy, patients continue to receive oral bafetinib twice daily in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days and then every 8 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have radiographic findings consistent with either:

  * Recurrent high-grade glioma, or
  * Metastatic disease to the brain that has progressed after treatment with whole brain radiation therapy or stereotactic radiosurgery; patients who have a resectable brain metastasis as the only site of disease (i.e., no evidence of systemic disease), are not eligible to participate
* Patients who are in need of a surgical debulking or a stereotactic biopsy for the purpose of diagnosis or differentiating between tumor progression versus treatment-induced effects following radiation therapy +/- chemotherapy will be eligible to participate in the microdialysis part of the study prior to beginning cycle 1 of bafetinib if the study neurosurgeon thinks there is a likelihood of being able to place the microdialysis catheter into residual tumor (enhancing brain tissue)
* Patients who choose not to participate in the microdialysis part of the study may enroll in the study and start treatment at cycle 1 of bafetinib
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for 3 months following duration of study participation; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately
* Patients must have a Karnofsky Performance Status (KPS) >= 60%
* If corticosteroids are required for controlling cerebral edema, patients must be on a stable dose for at least 1 week prior to enrollment
* Patients must not be taking any hepatic enzyme-inducing anticonvulsants (phenytoin, carbamazepine, phenobarbital, primidone, oxcarbazepine) for at least 2 weeks prior to enrollment
* Absolute neutrophil count >= 1500 cells/mm^3
* Platelet count >= 100,000 cells/mm^3
* Total bilirubin =< 2.0 mg/dl
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) =< 3 times the institutional upper limit of normal
* Alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) =< 3 times the institutional upper limit of normal
* Serum creatinine =< 1.5 x the institutional upper limit of normal
* QTc interval < 480 msec on electrocardiogram (ECG)
* All subjects must have the ability to understand and the willingness to sign a written informed consent
* Patients must have recovered from any toxicity of prior therapies (including brain radiation); an interval of at least 6 weeks must have elapsed since the completion of a nitrosourea-containing chemotherapy regimen; patients who have undergone a recent craniotomy cannot begin bafetinib until at least 2 weeks after the surgery

Exclusion Criteria:

* Patients who are currently receiving chemotherapy or are enrolled in another treatment clinical trial
* Patients with a coagulopathy or bleeding disorder
* Patients on anticoagulant drug therapy or medications that inhibit platelet function, such as ibuprofen or other non-steroidal anti-inflammatory drugs
* Clinically evident congestive heart failure > class II of the New York Heart Association (NYHA) guidelines
* Clinically significant cardiac arrhythmias
* Patients taking a drug that can prolong the QT interval; if a potential study patient is taking one of the prohibited drugs but s/he can safely stop it, then a washout period of >= 7 days is required prior to starting bafetinib
* History or signs of active coronary artery disease with or without angina pectoris
* Patients who have a serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol or may not be able to comply with the safety monitoring requirements of the study
* Human immunodeficiency virus (HIV)-positive patients receiving anti-retroviral therapy are excluded from the study due to the possibility of pharmacokinetic (PK) interactions with bafetinib; however, patients will not be routinely screened for HIV
* Female patients who are pregnant or breast-feeding
* Active, clinically significant serious infection requiring treatment with antibiotics, anti-virals or anti-fungals
* Patients who have not recovered from the toxicities of prior chemotherapy or radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Area-under-the-concentration-time-curve (AUC) of bafetinib in dialysate | every hour for 24 hours after first dose of bafetinib
Peak concentration (Cmax) of bafetinib in dialysate | every hour for 24 hours after first dose of bafetinib
AUC of bafetinib in plasma | 1, 2, 3, 4, 6, 8, and 12 hours after the first dose of bafetinib and then 1, 2, 3, 4, 6, 8, and 12 hours after the second dose of bafetinib
Cmax of bafetinib in plasma | 1, 2, 3, 4, 6, 8, and 12 hours after the first dose of bafetinib and then 1, 2, 3, 4, 6, 8, and 12 hours after the second dose of bafetinib

SECONDARY OUTCOMES:
Determination of adverse events associated with bafetinib in patient with recurrent malignant brain tumors | 30 days after last dose of bafetinib
Response rate in patients with malignant brain tumors treated with bafetinib | 30 days after last dose of bafetinib
Progression-free survival in patients with malignant brain tumors treated with bafetinib | 1 year after last dose of bafetinib
Overall survival in patients with malignant brain tumors treated with bafetinib | 2 years after last dose of bafetinib
Assessment for expression of Lyn and Fyn kinases and phosphorylation status in pre-treatment tumor samples. | Pre-treatment tumor samples

CONTACTS AND LOCATIONS:
Overall Officials: Jana Portnow, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - South Pasadena Cancer Center, South Pasadena, California

REFERENCES:
- [Derived] Portnow J, Badie B, Markel S, Liu A, D'Apuzzo M, Frankel P, Jandial R, Synold TW. A neuropharmacokinetic assessment of bafetinib, a second generation dual BCR-Abl/Lyn tyrosine kinase inhibitor, in patients with recurrent high-grade gliomas. Eur J Cancer. 2013 May;49(7):1634-40. doi: 10.1016/j.ejca.2013.01.001. Epub 2013 Feb 4. PMID 23380277